CLINICAL TRIAL: NCT01497132
Title: Effects of Vitamin D on Beta Cell Function and Insulin Sensitivity in Pre-diabetes and Diabetes Mellitus Type 2 - EVIDENS
Brief Title: Effects of Vitamin D on Beta Cell Function and Insulin Sensitivity in Pre-diabetes and Diabetes Mellitus Type 2
Acronym: EVIDENS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Henrik Wagner, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DvitamininDM2_v1_110815; 2010-024487-18 (EudraCT Number)
Record Dates: First submitted 2011-12-20; First posted 2011-12-22 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-09

CONDITIONS: Diabetes Mellitus, Type 2; Glucose Intolerance; Vitamin D Deficiency
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Intolerance; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D3 (Experimental)
  Interventions: Drug: Vitamin D3
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin D3 — Oral drops 30000 IU weekly
  Other Names: Vigantol oil
  Arms: Vitamin D3
Drug: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate if treatment with vitamin D increase beta cell function and insulin sensitivity in subjects with pre-diabetes or newly diagnosed diabetes mellitus type 2.

ELIGIBILITY:
Inclusion Criteria:

* Meeting criteria for IFG, IGT, IFG+IGT or diabetes mellitus at OGTT.
* BMI ≤ 32 kg/m2.
* HbA1c ≤ 7.0 % (MonoS) or ≤ 63 mmol/mol (IFCC).
* Fasting plasma glucose < 9 mmol/l
* S-25-OH-vitamin D3 < 75 nmol/l.

Exclusion Criteria:

* Treatment with any vitamin D preparation.
* Regular sun-bathing in solarium.
* Hypercalcemia at screening, defined as free s-calcium > 1.35 mmol/l.
* Hyperphosphatemia at screening, defined as s-phosphate > 1.5 mmol/l.
* Sarcoidosis or other granulomatous disease.
* Treatment with phenytoin, barbiturates, rifampicin, isoniazid, cardiac glycosides, orlistat or colestyramin.
* Impaired hepatic function.
* Impaired renal function
* Cardiac disease defined as:

  * Unstable angina pectoris
  * Myocardial infarction within the last 6 months
  * Congestive heart failure NYHA class III and IV
* Cerebral stroke within the last 6 months.
* Anti-diabetic medication of any kind.
* Females of childbearing potential who are pregnant, breast-feeding or intend to become pregnant or are not using adequate contraceptive methods.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Beta cell function | 8 weeks
  Assessed by hyperglycemic clamp investigation

SECONDARY OUTCOMES:
Insulin sensitivity | 8 weeks
  Assessed by hyperglycemic clamp investigation
Glucose tolerance | 8 weeks
  Assessed by OGTT
Hypercalcemia | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Wagner, M.D, Principal Investigator — Karolinska Institutet
Locations (1):
- Dpt of Endocrinology, Karolinska University Hospital, Stockholm, Stockholm County, Sweden

REFERENCES:
- [Derived] Wagner H, Alvarsson M, Mannheimer B, Degerblad M, Ostenson CG. No Effect of High-Dose Vitamin D Treatment on beta-Cell Function, Insulin Sensitivity, or Glucose Homeostasis in Subjects With Abnormal Glucose Tolerance: A Randomized Clinical Trial. Diabetes Care. 2016 Mar;39(3):345-52. doi: 10.2337/dc15-1057. Epub 2016 Jan 19. PMID 26786573
- [Derived] Mannheimer B, Wagner H, Ostenson CG, Diczfalusy U. No impact of vitamin D on the CYP3A biomarker 4beta-hydroxycholesterol in patients with abnormal glucose regulation. PLoS One. 2015 Apr 2;10(4):e0121984. doi: 10.1371/journal.pone.0121984. eCollection 2015. PMID 25835492